CLINICAL TRIAL: NCT04809623
Title: A Randomized, Blinded, Placebo-Controlled, Phase 1b Study of GS-5718 in Subjects With Cutaneous Lupus Erythematosus (CLE)
Brief Title: Study of Edecesertib in Participants With Cutaneous Lupus Erythematosus (CLE)
Acronym: LYNX
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision to terminate study.
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-497-5888; 2021-000204-38 (EudraCT Number)
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Results first posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2023-10

CONDITIONS: Cutaneous Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Edecesertib (Experimental): Participants continuing their standard of care therapy will receive edecesertib at a dose of 115 mg orally once daily for up to 4 weeks.
  Interventions: Drug: Edecesertib; Drug: Standard of Care
- Placebo (Experimental): Participants continuing their standard of care therapy will receive placebo to match edecesertib orally once daily for up to 4 weeks.
  Interventions: Drug: Placebo; Drug: Standard of Care

INTERVENTIONS:
Drug: Edecesertib — Tablets administered orally
  Other Names: GS-5718
  Arms: Edecesertib
Drug: Placebo — Placebo to match edecesertib tablets administered orally
  Arms: Placebo
Drug: Standard of Care — Immunosuppressive/immunomodulatory agents including but not limited to antimalarials (i.e. hydroxychloroquine), methotrexate, azathioprine and corticosteroids (i.e. prednisone)

SUMMARY:
The primary objective of this study is to evaluate the safety and tolerability of edecesertib (formerly GS-5718) in participants with cutaneous lupus erythematosus (CLE) with or without systemic lupus erythematosus (SLE).

ELIGIBILITY:
Key Inclusion Criteria:

* Either fulfill the European League Against Rheumatism (EULAR)/ American College of Rheumatology(ACR) 2019 classification criteria for systemic lupus erythematosus (SLE) or have biopsy-proven cutaneous lupus erythematosus (CLE).
* Must have active acute cutaneous lupus erythematosus (ACLE)/ subacute cutaneous lupus erythematosus (SCLE); individuals with mixed skin presentations of lupus skin disease (including DLE) are allowed to enter.
* CLE Disease Area and Severity Index (CLASI) activity score of ≥ 6 during screening and Day 1, excluding the alopecia component.
* Presence of at least 1 representative lupus skin lesion amenable to punch biopsy and willingness to undergo skin biopsy at 2 time points.
* Protocol-permitted nonbiologic immunosuppressive/immunomodulatory agents for the treatment of CLE/SLE (eg, antimalarials, methotrexate (MTX), or other conventional synthetic disease-modifying antirheumatic drug (csDMARDs)) must maintain stable dose(s) for ≥ 60 days prior to randomization through Week 4 of the study.

Key Exclusion Criteria:

* Dermatologic disease other than cutaneous manifestations of SLE or CLE that may interfere with assessment of lupus-specific skin lesions.
* Ongoing or active clinically significant bacterial, fungal or viral infection.
* History of or positive for human immunodeficiency virus, hepatitis C virus, or hepatitis B virus.
* Uncontrolled health conditions including highly active SLE (e.g. lupus nephritis, neuropsychiatric SLE, vasculitis etc.).
* History of malignancy.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (5):
- United States (5):
  - Wallace Rheumatic Studies Center, LLC, Beverly Hills, California
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Dawes Fretzin Clincial Research Group, LLC, Indianapolis, Indiana
  - DJL Clinical Research, PLLC, Charlotte, North Carolina
  - Metroplex Clinical Research Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study?nctid=NCT04809623

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at sites in the United States.
Pre-assignment Details: 7 participants were screened.
Groups:
- Edecesertib: Participants received edecesertib at a dose of 115 mg orally in form of tablets once daily for up to 4 weeks. The participants continued their standard of care therapy.
- Placebo: Participants received placebo to match edecesertib orally in form of tablets once daily for up to 4 weeks. The participants continued their standard of care therapy.
Period: Overall Study
Arm/Group | Edecesertib | Placebo
Started | 2 | 1
Completed | 1 | 1
Not Completed | 1 | 0
Not completed — Study Terminated by Sponsor | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Edecesertib | Placebo | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — Data not reported for participant confidentiality reasons. | NA (NA) — Data not reported for participant confidentiality reasons. | NA (NA) — Data not reported for participant confidentiality reasons.
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | NA — Data not reported for participant confidentiality reasons. | NA — Data not reported for participant confidentiality reasons. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Data not reported for participant confidentiality reasons. | NA — Data not reported for participant confidentiality reasons. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race/Ethnicity, Customized [Count of Participants; unit: Participants] | NA — Data not reported for participant confidentiality reasons. | NA — Data not reported for participant confidentiality reasons. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced Treatment-emergent Adverse Events
Description: Treatment-emergent Adverse Events (TEAEs) were defined as AEs with onset dates on or after the study treatment start date and no later than 28 days after the permanent discontinuation of the study treatment and/or the AEs that led to premature discontinuation of study treatments.
Time Frame: First dose date up to 4 weeks plus 28 days
Population: No data was reported for adverse events due to low number of participants in both Edicescertib and Placebo arms, in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Edecesertib | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Percentage of Participants Who Experienced Treatment-emergent Laboratory Abnormalities
Description: A treatment-emergent laboratory abnormality was defined as an increase of at least 1 abnormality grade from baseline and occurring after the first dose of study drug and within 28 days after last study drug administration.
Time Frame: First dose date up to 4 weeks plus 28 days
Population: as for outcome 1
Arm/Group | Edecesertib | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Pharmacokinetic (PK) Parameter: AUCtau of Edecesertib
Description: AUCtau is defined as the area under the concentration versus time curve over the dosing interval.
Time Frame: Predose and up to 6 hours postdose at Week 4
Population: Data not reported for participant confidentiality reasons.
Arm/Group | Edecesertib
Number analyzed (Participants) | 0

4. Secondary Outcome: Pharmacokinetic (PK) Parameter: Cmax of Edecesertib
Description: Cmax is defined as the maximum observed concentration of drug.
Time Frame: Predose and up to 6 hours postdose at Week 4
Population: Data not reported for participant confidentiality reasons.
Arm/Group | Edecesertib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose date up to 4 weeks plus 28 days All-Cause Mortality: First dose date up to approximately 10 weeks
Description: No data was reported for adverse events due to low number of participants in both Edicescertib and Placebo arms, in order to protect and maintain participant privacy/confidentiality.
Arm/Group | Edecesertib | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years.

DOCUMENTS (2):
  • Study Protocol (2021-07-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT04809623/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-13): https://cdn.clinicaltrials.gov/large-docs/23/NCT04809623/SAP_001.pdf